CLINICAL TRIAL: NCT01559363
Title: A Phase 1b/2a, Safety, Pharmacokinetic and Dose-Escalation Study of KD019 (Tesevatinib) in Subjects With Autosomal Dominant Polycystic Kidney Disease (ADPKD)
Brief Title: A Safety, Pharmacokinetic & Dose-Escalation Study of KD019 in Subjects With Autosomal Dominant Polycystic Kidney Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KD019-101; U1111-1279-2764 (Other: UTN); MAD17715 (Other: Sanofi study ID)
Record Dates: First submitted 2012-03-09; First posted 2012-03-21 (Estimated); Results first posted 2022-11-08 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Polycystic Kidney, Autosomal Dominant
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing (Experimental): Participants received tesevatinib 50 milligrams (mg) tablet orally once daily (QD) for 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum duration: up to 36 months).
  Interventions: Drug: Tesevatinib
- Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing (Experimental): Participants received tesevatinib 100 mg tablet orally QD for 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 36 months).
  Interventions: Drug: Tesevatinib
- Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing (Experimental): Participants received tesevatinib 150 mg tablet orally QD for 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 36 months).
  Interventions: Drug: Tesevatinib
- Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing (Experimental): Participants received tesevatinib 150 mg tablet orally bi-weekly in alternative dosing schedules on Monday and Thursday for initial 25 days. After initial 25 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 28 months).
  Interventions: Drug: Tesevatinib
- Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing (Experimental): Participants received tesevatinib 150 mg tablet orally tri-weekly in alternative dosing schedules on Monday, Wednesday and Friday for initial 26 days. After initial 26 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 28 months).
  Interventions: Drug: Tesevatinib
- Phase 2a: Safety in Larger Kidneys (SILK) Cohort: Tesevatinib 50 mg Once Daily Dosing (Experimental): Participants with autosomal dominant polycystic kidney disease (and Baseline estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 35 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) and less than or equal to (<=) 80 mL/min/1.73 m^2, and height-adjusted total kidney volume (htTKV) >=1000 mL were enrolled and received tesevatinib 50 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 28 months).
  Interventions: Drug: Tesevatinib

INTERVENTIONS:
Drug: Tesevatinib — Pharmaceutical form: Tablets Route of administration: Oral
  Other Names: XL647 and KD019

SUMMARY:
The primary objective of this study Phase 1b was to determine the safety, plasma pharmacokinetics, and maximum tolerated dose (MTD) of tesevatinib when administered to participants with autosomal dominant polycystic kidney disease (ADPKD).

The primary objective of this study Phase 2a was to evaluate the annualized change in glomerular filtration rate (GFR) in participants with ADPKD when treated with tesevatinib.

DETAILED DESCRIPTION:
Phase 1b:

* Primary objective was to determine the safety of tesevatinib.
* Dosing was for 28 days daily. After the 28-day treatment period, participants would, at the discretion of the investigator, continue to receive study treatment for 24 months from their first dose or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision. Participants might continue beyond 24 months at the discretion of the investigator after consultation with the medical monitor.
* All participants received active tesevatinib study drug.
* Tesevatinib is an oral once daily tablet. Tablets were 50 milligrams (mg), 100 mg and 150 mg in strength. Participants were enrolled into three sequential dosing cohort levels (50 mg, 100 mg and 150 mg.). Participants in Phase 1b had their dose increased or decreased to the maximum tolerated dose (MTD).
* Study participants had magnetic resonance imaging (MRI) of the abdomen (kidneys) at Screening and 6 months thereafter to explore effects of KD019.
* Echocardiogram was performed at Screening, Day 28, months 3 and 6 and every 6 months thereafter.

Phase 2a:

* Primary objective was to compare the annualized change in GFR in participants with ADPKD when treated with tesevatinib.
* Two alternate dosing schedules were explored to determine if they were more tolerable than daily dosing when used chronically in participants with ADPKD.
* Participants received study treatment for 24 months from their first dose or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision. Participants continued beyond 24 months at the discretion of the investigator after consultation with the sponsor.
* All participants received active tesevatinib study drug.
* Tablets were 50 mg, 100 mg, and 150 mg in strength.
* Study participants had MRI of the abdomen (kidneys) at Screening and Month 6 visit and every 6 months after to explore effects of tesevatinib.
* Echocardiogram was performed at Screening, Day 28, and Months 3 and 6 and 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* The participant had a confirmed diagnosis of ADPKD.
* The participant had a GFR >=35 mL/min/1.73m^2.
* Cysts must be at least 1 centimeter in size.
* Adequate bone marrow, kidney, and liver function.
* Must agree to use two forms of birth control for those of child bearing potential.
* Normal amylase and lipase levels.
* The participant had a htTKV >= 1000 mL (htTKV was calculated using total kidney volume obtained from magnetic resonance imaging divided by height in meters).

Exclusion Criteria:

* The participant has had a previous partial or total nephrectomy.
* The participant had tuberous sclerosis, Hippel-Lindau disease, or acquired cystic disease.
* The participant had congenital absence of one kidney and/or need for dialysis.
* Presence of renal or hepatic calculi (stones) causing symptoms.
* The participant had received any investigational therapy within 30 days prior to study entry.
* Active treatment (within 4 weeks of study entry) for urinary tract infection.
* Participant was known to be immunocompromised.
* Participant was pregnant or nursing.
* History of pericardial effusion or presence of pericardial effusion on screening echocardiogram
* Uncontrolled hypertension.
* History of pancreatitis or had known risk factors for pancreatitis.
* Participant had received EGFR inhibitor at any time.
* The participant was aphakic due to previous cataract surgery or congenital anomaly.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2012-10-11 (Actual); Primary Completion 2019-02-08 (Actual); Study Completion 2019-02-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado Denver, Denver, Colorado
  - University of Kansas Medical Center, Kansas City, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New York University School of Medicine, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Clinical Advancement Center, PLLC, San Antonio, Texas
  - University of Virginia - Nephrology Clinical Research Center, Charlottesville, Virginia
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 11 active sites in the United States. A total of 126 participants were screened between 11 October 2012 and 07 March 2017, of which 69 participants were enrolled and treated.
Pre-assignment Details: Study consisted of 2 parts: Phase 1b with three sequential dosing cohort levels (50 milligrams [mg], 100 mg and 150 mg) and Phase 2a with two alternate dosing schedules cohorts (150 mg biweekly and triweekly) and one safety in larger kidneys (SILK) cohort.
Groups:
- Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing: Participants received tesevatinib 50 mg tablet orally once daily (QD) for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 36 months).
- Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing: Participants received tesevatinib 100 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 36 months).
- Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing: Participants received tesevatinib 150 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 36 months).
- Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing: Participants with autosomal dominant polycystic kidney disease (ADPKD) and Baseline estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 35 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) and less than or equal to (<=) 80 mL/min/1.73 m^2, and height-adjusted total kidney volume (htTKV) >=1000 mL were enrolled and received tesevatinib 50 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 28 months).
Period: Phase 1b: Up to 36 Months
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
Started | 24 | 8 | 5 | 0 | 0 | 0
Completed | 18 | 5 | 3 | 0 | 0 | 0
Not Completed | 6 | 3 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Investigator decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse event or Serious adverse event | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Unspecified reason | 0 | 1 | 0 | 0 | 0 | 0
Period: Phase 2a: Up to 28 Months
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
Started | 0 | 0 | 0 | 10 (Phase 2b and Phase 1b were separate populations.) | 14 (Phase 2b and Phase 1b were separate populations.) | 8 (Phase 2b and Phase 1b were separate populations.)
Completed | 0 | 0 | 0 | 8 | 13 | 8
Not Completed | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Adverse event or Serious adverse event | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Unspecified reason | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population which included all participants who receive at least 1 dose of tesevatinib.
Groups:
- Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing: Participants received tesevatinib 50 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum duration: up to 36 months).
- Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing: Participants with ADPKD and Baseline eGFR >=35 mL/min/1.73 m^2 and <=80 mL/min/1.73 m^2, and htTKV >=1000 mL were enrolled and received tesevatinib 50 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 28 months).
- Total: Total of all reporting groups
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing | Total
Number analyzed (Participants) | 24 | 8 | 5 | 10 | 14 | 8 | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (9.1) | 36.6 (7.4) | 42.6 (4.4) | 34.9 (11.3) | 37.7 (11.1) | 52.1 (9.5) | 39.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 3 | 3 | 6 | 10 | 3 | 40
  Male | 9 | 5 | 2 | 4 | 4 | 5 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 0 | 0 | 0 | 0 | 0 | 3
  White | 20 | 8 | 5 | 8 | 14 | 7 | 62
  Black or African American | 1 | 0 | 0 | 2 | 0 | 0 | 3
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAE)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal product and which did not necessarily had to have a causal relationship with the treatment. An SAE was any untoward medical occurrence at any dose that: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were AEs that developed or worsened or became serious from the first dose (Day 1) of the study drug until 30 days after the last dose of study drug.
Time Frame: From Baseline (Day 1) until 30 days after the last dose of study drug (maximum duration: up to 37 months)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 24 | 8 | 5
Participants
  TEAEs | 24 | 8 | 5
  SAE | 1 | 0 | 0

2. Primary Outcome: Phase 1b: Pharmacokinetics (PK): Plasma Concentrations of Tesevatinib 100 mg and 150 mg
Description: Plasma concentrations of tesevatinib was analyzed using non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: Analysis was performed on PK Population which consisted of all participants who received at least one dose of tesevatinib 100 mg (in Phase 1b: Cohort 2) and 150 mg (in Phase 1b: Cohort 3) and had quantifiable PK data available. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 8 | 5
nanograms per milliliter (ng/mL)
  Day 1: Pre-dose | 0 (0) | 0 (0)
  Day 1: 1 hour post-dose | 4.39 (2.78) | 8.41 (5.84)
  Day 1: 2 hours post-dose | 10.1 (10.2) | 18.6 (12.0)
  Day 1: 4 hours post-dose | 21.1 (14.8) | 33.1 (8.24)
  Day 1: 8 hours post-dose | 25.4 (12.1) | 44.3 (7.50)
  Day 1: 24 hours post-dose | 21.9 (9.69) | 35.5 (7.10)
  Day 14: Pre-dose | 90.3 (29.1) | 164 (45.4)
  Day 14: 1 hour post-dose | 94.0 (26.9) | 160 (37.2)
  Day 14: 2 hours post-dose | 103 (29.4) | 180 (47.3)
  Day 14: 4 hours post-dose | 111 (39.7) | 204 (66.8)
  Day 14: 24 hours post-dose: number analyzed (Participants) | 7 | 5
  Day 14: 24 hours post-dose | 91.1 (28.9) | 150 (37.0)

3. Primary Outcome: Phase 1b: Pharmacokinetics: Plasma Concentrations of Tesevatinib 50 mg
Description: Plasma concentrations of tesevatinib was analyzed using non-compartmental analysis.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: Analysis was performed on PK Population which consisted of all participants who received at least one dose of tesevatinib 50 mg in Phase 1b and had quantifiable PK data available. Here, overall number of participants analyzed = participants evaluable for this outcome measure (OM) and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 23
ng/mL
  Day 1: Pre-dose | 0 (0)
  Day 1: 1 hour post-dose | 2.20 (2.06)
  Day 1: 2 hours post-dose: number analyzed (Participants) | 22
  Day 1: 2 hours post-dose | 5.22 (3.58)
  Day 1: 4 hours post-dose | 10.4 (4.77)
  Day 1: 8 hours post-dose: number analyzed (Participants) | 22
  Day 1: 8 hours post-dose | 12.1 (5.74)
  Day 1: 24 hours post-dose: number analyzed (Participants) | 22
  Day 1: 24 hours post-dose | 13.6 (4.18)
  Day 14: Pre-dose: number analyzed (Participants) | 21
  Day 14: Pre-dose | 54.4 (20.5)
  Day 14: 1 hour post-dose: number analyzed (Participants) | 20
  Day 14: 1 hour post-dose | 56.8 (22.3)
  Day 14: 2 hours post-dose: number analyzed (Participants) | 20
  Day 14: 2 hours post-dose | 58.5 (23.2)
  Day 14: 4 hours post-dose: number analyzed (Participants) | 20
  Day 14: 4 hours post-dose | 63.2 (23.3)
  Day 14: 24 hours post-dose: number analyzed (Participants) | 20
  Day 14: 24 hours post-dose | 55.8 (19.1)

4. Primary Outcome: Phase 1b: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of Tesevatinib 100 mg and 150 mg
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: Analysis was performed on PK Population.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 8 | 5
ng/mL
  Day 1 | 27.5 (12.2) | 44.3 (7.50)
  Day 14 | 116 (31.8) | 205 (65.4)

5. Primary Outcome: Phase 1b: Pharmacokinetics: Maximum Observed Plasma Concentration of Tesevatinib 50 mg
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: Analysis was performed on PK Population. Here, overall number of participants analyzed = participants evaluable for this OM and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 23
ng/mL
  Day 1 | 14.5 (5.34)
  Day 14: number analyzed (Participants) | 20
  Day 14 | 65.9 (24.8)

6. Primary Outcome: Phase 1b: Pharmacokinetics: Time of the Maximum Observed Plasma Concentration (Tmax) of Tesevatinib 100 mg and 150 mg
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: Analysis was performed on PK Population.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 8 | 5
hours
  Day 1 | 10.9 (8.09) | 7.99 (0.0434)
  Day 14 | 6.25 (7.01) | 3.59 (0.891)

7. Primary Outcome: Phase 1b: Pharmacokinetics: Time of the Maximum Observed Plasma Concentration of Tesevatinib 50 mg
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 23
hours
  Day 1 | 16.4 (8.86)
  Day 14: number analyzed (Participants) | 20
  Day 14 | 5.33 (6.34)

8. Primary Outcome: Phase 1b: Pharmacokinetics: Time of the Last Quantifiable Plasma Concentration (Tlast) of Tesevatinib 100 mg and 150 mg
Description: Tlast was defined as time to reach last quantifiable plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: Analysis was performed on PK Population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- Phase 1b: Cohort 3: Tesevatinib 150 mg: Participants received tesevatinib 150 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 36 months).
Arm/Group | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg
Number analyzed (Participants) | 8 | 5
hours
  Day 1 | 23.9 (0.264) | 23.9 (0.132)
  Day 14: number analyzed (Participants) | 7 | 5
  Day 14 | 23.5 (0.606) | 23.9 (0.154)

9. Primary Outcome: Phase 1b: Pharmacokinetics: Time of the Last Quantifiable Plasma Concentration of Tesevatinib 50 mg
Description: Tlast was defined as time to reach last quantifiable plasma concentration.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 22
hours
  Day 1 | 23.9 (0.177)
  Day 14: number analyzed (Participants) | 20
  Day 14 | 23.9 (0.266)

10. Primary Outcome: Phase 1b: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration (AUC0-t) of Tesevatinib 100 mg and 150 mg
Description: AUC0-last was defined as area under the concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration (tlast).
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hour*nanograms per milliliter (hr*ng/mL)
Arm/Group | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 8 | 5
hour*nanograms per milliliter (hr*ng/mL)
  Day 1 | 508 (247) | 853 (130)
  Day 14: number analyzed (Participants) | 7 | 5
  Day 14 | 2280 (741) | 4200 (1180)

11. Primary Outcome: Phase 1b: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of Last Quantifiable Concentration of Tesevatinib 50 mg
Description: as for outcome 10
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 21
hr*ng/mL
  Day 1 | 272 (99.9)
  Day 14: number analyzed (Participants) | 20
  Day 14 | 1410 (485)

12. Primary Outcome: Phase 1b: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time Zero to 24 Hours Post-dose (AUC0-24) of Tesevatinib 100 mg and 150 mg
Description: AUC0-24 was defined as area under the plasma concentration versus time curve of study drug from time 0 to 24 hours post-dose.
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 8 | 5
hr*ng/mL
  Day 1 | 507 (246) | 853 (129)
  Day 14: number analyzed (Participants) | 6 | 5
  Day 14 | 2700 (750) | 4200 (1180)

13. Primary Outcome: Phase 1b: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Post-dose of Tesevatinib 50 mg
Description: as for outcome 12
Time Frame: Pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and pre-dose, 1, 2, 4, and 24 hours post-dose on Day 14
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 21
hr*ng/mL
  Day 1 | 272 (99.8)
  Day 14: number analyzed (Participants) | 18
  Day 14 | 1430 (498)

14. Primary Outcome: Phase 1b: Pharmacokinetics: Trough Plasma Concentrations (Ctrough) of Tesevatinib 100 mg and 500 mg
Description: Ctrough was the plasma concentration observed at the time immediately before (pre-dose) study drug administration.
Time Frame: Pre-dose on Days 7, 14, 21, 28 and Months 2, 3, 4, 5 and 6
Population: as for outcome 8
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 8 | 5
ng/mL
  Day 7: Pre-dose: number analyzed (Participants) | 8 | 4
  Day 7: Pre-dose | 72.7 [52.0 to 108] | 143 [75.5 to 173]
  Day 14: Pre-dose | 90.3 [52.8 to 131] | 164 [105 to 213]
  Day 21: Pre-dose | 88.1 [5.74 to 122] | 155 [17.5 to 230]
  Day 28: Pre-dose: number analyzed (Participants) | 8 | 4
  Day 28: Pre-dose | 93.7 [22.9 to 135] | 180 [137 to 207]
  Month 2: Pre-dose: number analyzed (Participants) | 8 | 1
  Month 2: Pre-dose | 87.0 [17.1 to 142] | 107 [107 to 107]
  Month 3: Pre-dose: number analyzed (Participants) | 6 | 2
  Month 3: Pre-dose | 113 [80.3 to 152] | 130.25 [96.5 to 164]
  Month 4: Pre-dose: number analyzed (Participants) | 6 | 1
  Month 4: Pre-dose | 128 [83.4 to 173] | 121 [121 to 121]
  Month 5: Pre-dose: number analyzed (Participants) | 5 | 2
  Month 5: Pre-dose | 89.0 [66.4 to 116] | 227.5 [122 to 333]
  Month 6: Pre-dose: number analyzed (Participants) | 5 | 2
  Month 6: Pre-dose | 84.7 [63.2 to 112] | 119 [110 to 128]

15. Primary Outcome: Phase 1b: Pharmacokinetics: Trough Plasma Concentrations of Tesevatinib 50 mg
Description: Ctrough was the plasma concentration observed at the time immediately before study drug administration.
Time Frame: Pre-dose on Days 7, 14, 21, 28 and Months 2, 3, 4, 5 and 6
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 22
ng/mL
  Day 7: Pre-dose | 45.4 (14.8)
  Day 14: Pre-dose: number analyzed (Participants) | 21
  Day 14: Pre-dose | 54.4 (20.5)
  Day 21: Pre-dose: number analyzed (Participants) | 19
  Day 21: Pre-dose | 59.9 (23.8)
  Day 28: Pre-dose: number analyzed (Participants) | 20
  Day 28: Pre-dose | 59.5 (26.7)
  Month 2: Pre-dose: number analyzed (Participants) | 18
  Month 2: Pre-dose | 54.9 (24.5)
  Month 3: Pre-dose: number analyzed (Participants) | 17
  Month 3: Pre-dose | 50.0 (21.8)
  Month 4: Pre-dose: number analyzed (Participants) | 16
  Month 4: Pre-dose | 45.5 (17.4)
  Month 5: Pre-dose: number analyzed (Participants) | 15
  Month 5: Pre-dose | 46.5 (16.3)
  Month 6: Pre-dose: number analyzed (Participants) | 15
  Month 6: Pre-dose | 44.8 (17.9)

16. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) of Tesevatinib
Description: The MTD was determined based on dose-limiting toxicities (DLTs) occurring in the first 28 days of study treatment. Any toxicity that the Investigator and the Sponsor deemed to be dose-limiting, regardless of the grade, was considered as DLT.
Time Frame: Cycle 1 (Up to 28 days)
Population: Analysis was performed on safety population. Data for this OM was not planned to be collected and analyzed for Phase 2a participants as pre specified in protocol.
Measure: Number; unit: milligrams
Groups:
- Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing: Participants received tesevatinib 50 mg tablet orally QD for initial 28 days. After initial 28 days treatment, at the investigator's discretion, participants continued to receive tesevatinib for a total of 24 months (since treatment initiation) or until the development of unacceptable toxicity, noncompliance, or withdrawal of consent by the participant, or investigator decision (maximum exposure duration: up to 36 months).
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing
Number analyzed (Participants) | 24 | 8 | 5
milligrams | 100 | 100 | 100

17. Primary Outcome: Phase 2a: Annualized Percent Change From Baseline in Estimated Glomerular Filtration Rate (eGFR)
Description: eGFR: measures kidney function based on serum creatinine (Scr) and cystatin C (Scys). Annualized change in eGFR was calculated as: percent change from Baseline divided by total duration in days*365.25. eGFR was estimated using 3 formulas and is reported separately for each formula: 1) 4-variable modification of diet in renal disease (MDRD-4) : Black/African-American males:175*(Creatinine [Cr]^-1.154)*(Age^-0.203)*1.212, other males:175*(Cr^-1.154)*(Age^-0.203), females: male equation*0.742.; 2) cystatin C-based chronic kidney disease (CKD) epidemiology (EPI) (CKD-EPI2012cys) equation: based on Scyc levels, for males if <=0.8: 133*(Scys/0.8)^0.499*0.996^age, if >0.8: 133*(Scys/0.8)^-1.238*0.996^age; for female: male equation*0.932., 3) Scr- and Scys-based CKD-EPI (CKD EPI2012Scr-cys) equation: 135*(Scr/0.9)^XX*(Scys/0.8)^XXX*0.995^age*(× 1.08, if black)- XX and XXX had variable values based on different values of Scr and Scys.
Time Frame: Baseline (Day 1), Months 6, 12, 18, 24 and at end of study (i.e., anytime up to 37 months)
Population: Analyzed on modified intent-to-treat (mITT) population which included all participants who completed 25 days (Phase 2a participants in the Monday/Thursday dosing cohort), 26 days (Phase 2a participants in the Monday/Wednesday/Friday dosing cohort), and 28 days (SILK Cohort). Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for Phase 1b participants as pre specified in protocol.
Measure: Mean (Standard Deviation); unit: percent change/participant-year
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 10 | 12 | 8
percent change/participant-year
  Month 6: MDRD-4: number analyzed (Participants) | 8 | 11 | 8
  Month 6: MDRD-4 | -0.125 (0.3236) | -0.150 (0.1515) | -0.195 (0.1851)
  Month 6: CKD-EPI2012cys: number analyzed (Participants) | 8 | 11 | 8
  Month 6: CKD-EPI2012cys | 0.069 (0.2150) | 0.125 (0.1795) | 0.131 (0.2310)
  Month 6: CKD-EPI2012Scr-cys: number analyzed (Participants) | 8 | 11 | 8
  Month 6: CKD-EPI2012Scr-cys | -0.031 (0.1522) | -0.009 (0.1277) | -0.043 (0.1341)
  Month 12: MDRD-4: number analyzed (Participants) | 8 | 11 | 7
  Month 12: MDRD-4 | -0.096 (0.1177) | -0.103 (0.1222) | -0.173 (0.0515)
  Month 12: CKD-EPI2012cys: number analyzed (Participants) | 8 | 11 | 7
  Month 12: CKD-EPI2012cys | 0.040 (0.0644) | 0.031 (0.0696) | -0.037 (0.0966)
  Month 12: CKD-EPI2012Scr-cys: number analyzed (Participants) | 8 | 11 | 7
  Month 12: CKD-EPI2012Scr-cys | -0.028 (0.0721) | -0.040 (0.0861) | -0.113 (0.0565)
  Month 18: MDRD-4: number analyzed (Participants) | 7 | 11 | 7
  Month 18: MDRD-4 | -0.087 (0.0680) | -0.060 (0.0402) | -0.121 (0.1002)
  Month 18: CKD-EPI2012cys: number analyzed (Participants) | 7 | 11 | 7
  Month 18: CKD-EPI2012cys | 0.006 (0.0251) | 0.055 (0.0674) | 0.024 (0.1167)
  Month 18: CKD-EPI2012Scr-cys: number analyzed (Participants) | 7 | 11 | 7
  Month 18: CKD-EPI2012Scr-cys | -0.040 (0.0379) | 0.000 (0.0463) | -0.056 (0.1049)
  Month 24: MDRD-4: number analyzed (Participants) | 6 | 10 | 7
  Month 24: MDRD-4 | -0.010 (0.0657) | -0.049 (0.0500) | -0.077 (0.0752)
  Month 24: CKD-EPI2012cys: number analyzed (Participants) | 6 | 11 | 7
  Month 24: CKD-EPI2012cys | -0.000 (0.0245) | 0.029 (0.0388) | -0.017 (0.1081)
  Month 24: CKD-EPI2012Scr-cys: number analyzed (Participants) | 6 | 10 | 7
  Month 24: CKD-EPI2012Scr-cys | -0.008 (0.0240) | -0.015 (0.0251) | -0.051 (0.0734)
  End of study: MDRD-4: number analyzed (Participants) | 10 | 5 | 8
  End of study: MDRD-4 | -0.026 (0.2369) | -0.084 (0.1903) | -0.021 (0.0836)
  End of study: CKD-EPI2012cys: number analyzed (Participants) | 10 | 5 | 8
  End of study: CKD-EPI2012cys | 0.005 (0.0937) | 0.128 (0.2872) | -0.061 (0.0827)
  End of study: CKD-EPI2012Scr-cys: number analyzed (Participants) | 10 | 5 | 8
  End of study: CKD-EPI2012Scr-cys | -0.018 (0.1259) | 0.014 (0.0451) | -0.045 (0.0723)

18. Secondary Outcome: Phase 2a: Annualized Percent Change From Baseline in Height Adjusted Total Kidney Volume (htTKV) at Month 6, 12, 18, 24 and End of Study
Description: htTKV was calculated using total kidney volume obtained from magnetic resonance imaging (MRI) divided by height in meters. The annualized percent change from Baseline was calculated as the percent change from Baseline divided by total duration in days*365.25.
Time Frame: Baseline (Day 1), Months 6, 12, 18, 24 and at end of study (i.e., anytime up to 37 months)
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category. Data for this OM was not planned to be collected and analyzed for Phase 1b participants as pre specified in protocol.
Measure: Mean (Standard Deviation); unit: percent change/participant-year
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 10 | 12 | 8
percent change/participant-year
  Month 6: number analyzed (Participants) | 8 | 10 | 8
  Month 6 | 0.0696 (0.1161) | 0.0544 (0.1292) | 0.1570 (0.0943)
  Month 12: number analyzed (Participants) | 8 | 10 | 7
  Month 12 | 0.0503 (0.0758) | 0.0422 (0.0687) | 0.1145 (0.0722)
  Month 18: number analyzed (Participants) | 7 | 10 | 7
  Month 18 | 0.0632 (0.0512) | 0.0353 (0.0483) | 0.0841 (0.0277)
  Month 24: number analyzed (Participants) | 5 | 10 | 7
  Month 24 | 0.0702 (0.0517) | 0.0540 (0.0584) | 0.1080 (0.0536)
  End of study: number analyzed (Participants) | 1 | 5 | 1
  End of study | 0.0943 | 0.0517 (0.0327) | 0.0731

19. Secondary Outcome: Phase 2a: Annualized Percent Change From Baseline in the Reciprocal of Serum Creatinine at End of Study
Description: Reciprocal Creatinine was an indication for monitoring renal disease progression over time. The annualized percent change from Baseline was calculated as the percent change from Baseline divided by total duration in days*365.25.
Time Frame: Baseline (Day 1), at end of study (i.e., anytime up to 37 months)
Population: Analysis was performed on mITT Population. Data for this OM was not planned to be collected and analyzed for Phase 1b participants as pre specified in protocol.
Measure: Mean (Standard Deviation); unit: percent change per participant-year
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 10 | 12 | 8
percent change per participant-year | -8.2923 (29.0965) | -6.9630 (20.2475) | 4.0189 (20.0561)

20. Secondary Outcome: Phase 2a: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (TESAE)
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal product and which did not necessarily had to have a causal relationship with the treatment. An SAE was any untoward medical occurrence at any dose that: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were AEs that developed or worsened or became serious from the first dose (Day 1) of the study drug until 30 days after the last dose of study drug.
Time Frame: From Baseline (Day 1) until 30 days after the last dose of study drug (i.e., up to 29 months)
Population: Analysis was performed on safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 10 | 14 | 8
Participants
  TEAEs | 10 | 14 | 8
  SAEs | 1 | 0 | 1

21. Secondary Outcome: Phase 2a: Change From Baseline in Serum Creatinine Levels
Description: Serum creatinine levels indicated the renal function (normal or abnormal) over time.
Time Frame: Baseline, Day 1, 3, 7, 11, 12, 14, 21, 25, 26, 28, Month 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 16, 18, 20, 22, 24, and at end of study (i.e., anytime up to 37 months)
Population: Analysis was performed on safety population. Here, 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint. Data for this OM was not planned to be collected and analyzed for Phase 1b participants as pre specified in protocol.
Measure: Mean (Standard Deviation); unit: micromoles per liter
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
Number analyzed (Participants) | 10 | 14 | 8
micromoles per liter
  Day 1: number analyzed (Participants) | 0 | 0 | 2
  Day 1 |  |  | 35.5 (34.6)
  Day 3: number analyzed (Participants) | 0 | 0 | 4
  Day 3 |  |  | 9.8 (11.4)
  Day 7: number analyzed (Participants) | 0 | 0 | 8
  Day 7 |  |  | 11.1 (15.6)
  Day 11: number analyzed (Participants) | 10 | 0 | 0
  Day 11 | 4.5 (9.0) |  |
  Day 12: number analyzed (Participants) | 0 | 12 | 0
  Day 12 |  | 12.5 (8.5) |
  Day 14: number analyzed (Participants) | 0 | 0 | 8
  Day 14 |  |  | 8.3 (12.2)
  Day 21: number analyzed (Participants) | 0 | 0 | 8
  Day 21 |  |  | 14.9 (17.5)
  Day 25: number analyzed (Participants) | 10 | 0 | 0
  Day 25 | 5.3 (10.9) |  |
  Day 26: number analyzed (Participants) | 0 | 12 | 0
  Day 26 |  | 8.2 (6.4) |
  Day 28: number analyzed (Participants) | 0 | 0 | 8
  Day 28 |  |  | 14.9 (15.2)
  Month 2: number analyzed (Participants) | 9 | 12 | 7
  Month 2 | 9.6 (14.1) | 5.8 (7.3) | 7.4 (20.5)
  Month 3: number analyzed (Participants) | 9 | 12 | 8
  Month 3 | 8.4 (11.6) | 7.3 (8.6) | 10.8 (10.7)
  Month 4: number analyzed (Participants) | 8 | 12 | 8
  Month 4 | 10.6 (14.0) | 4.5 (12.0) | 14.6 (12.4)
  Month 5: number analyzed (Participants) | 8 | 10 | 7
  Month 5 | 4.4 (12.9) | 4.6 (6.9) | 7.1 (10.6)
  Month 6: number analyzed (Participants) | 8 | 11 | 8
  Month 6 | 5.4 (11.0) | 5.5 (5.6) | 10.4 (9.9)
  Month 7: number analyzed (Participants) | 7 | 10 | 8
  Month 7 | 9.6 (9.6) | 6.1 (6.0) | 24.9 (26.2)
  Month 8: number analyzed (Participants) | 8 | 11 | 8
  Month 8 | 11.4 (11.1) | 5.4 (6.7) | 9.4 (8.3)
  Month 9: number analyzed (Participants) | 8 | 11 | 7
  Month 9 | 10.6 (11.8) | 6.5 (7.7) | 12.0 (17.2)
  Month 10: number analyzed (Participants) | 8 | 10 | 7
  Month 10 | 7.5 (13.7) | 2.6 (7.8) | 14.6 (9.0)
  Month 11: number analyzed (Participants) | 8 | 11 | 7
  Month 11 | 12.1 (11.3) | 9.2 (9.5) | 13.3 (18.7)
  Month 12: number analyzed (Participants) | 8 | 11 | 7
  Month 12 | 8.6 (10.4) | 8.0 (9.8) | 20.7 (9.7)
  Month 13: number analyzed (Participants) | 0 | 0 | 1
  Month 13 |  |  | 0.0
  Month 14: number analyzed (Participants) | 8 | 11 | 7
  Month 14 | 6.1 (10.0) | 13.6 (9.8) | 13.3 (8.7)
  Month 16: number analyzed (Participants) | 7 | 11 | 7
  Month 16 | 11.7 (11.5) | 6.7 (7.2) | 15.6 (13.1)
  Month 18: number analyzed (Participants) | 7 | 11 | 7
  Month 18 | 11.4 (11.3) | 6.6 (4.2) | 21.6 (17.4)
  Month 20: number analyzed (Participants) | 6 | 10 | 7
  Month 20 | 5.7 (11.4) | 4.6 (9.1) | 12.3 (26.9)
  Month 22: number analyzed (Participants) | 6 | 11 | 7
  Month 22 | 6.7 (11.2) | 5.9 (10.3) | 12.3 (20.3)
  Month 24: number analyzed (Participants) | 6 | 10 | 7
  Month 24 | 2.8 (10.6) | 7.0 (7.0) | 18.0 (20.6)
  End of study: number analyzed (Participants) | 10 | 5 | 8
  End of study | 5.5 (10.1) | 3.6 (8.3) | 6.3 (17.4)

22. Secondary Outcome: Phase 2a: Pharmacokinetics: Plasma Concentrations of Tesevatinib 150 mg
Description: Plasma concentrations of tesevatinib was analyzed using non-compartmental analysis.
Time Frame: Bi-weekly: pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1 and Day 25; Tri-weekly: pre-dose, 1, 2, 4, 8, and 24 hours post-dose on Day 1; pre-dose, 1, 2, 4, and 24 hours post-dose on Day 12
Population: Analysis was performed on PK population. Here, overall number of participants analyzed = participants evaluable for this OM and 'number analyzed' = participants with available data for each specified category and '0' in the number analyzed field signifies that none of the participants were evaluable at the specified timepoint. Data for this OM was not planned to be collected and analyzed for Phase 2a SILK cohort participants.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing
Number analyzed (Participants) | 5 | 5
ng/mL
  Day 1: pre-dose | 0 (0) | 0 (0)
  Day 1: 1 hour post-dose | 14.8 (18.9) | 13.0 (11.2)
  Day 1: 2 hours post-dose | 21.7 (14.7) | 20.9 (12.7)
  Day 1: 4 hours post-dose | 46.0 (16.2) | 41.1 (25.4)
  Day 1: 8 hours post-dose | 55.0 (16.7) | 49.8 (19.9)
  Day 1: 24 hours post-dose: number analyzed (Participants) | 5 | 4
  Day 1: 24 hours post-dose | 45.4 (8.81) | 42.4 (13.0)
  Day 12: pre-dose: number analyzed (Participants) | 0 | 5
  Day 12: pre-dose |  | 53.7 (24.8)
  Day 12: 1 hour post-dose: number analyzed (Participants) | 0 | 5
  Day 12: 1 hour post-dose |  | 58.5 (21.1)
  Day 12: 2 hours post-dose: number analyzed (Participants) | 0 | 5
  Day 12: 2 hours post-dose |  | 70.1 (26.5)
  Day 12: 4 hours post-dose: number analyzed (Participants) | 0 | 5
  Day 12: 4 hours post-dose |  | 100 (42.6)
  Day 12: 24 hours post-dose: number analyzed (Participants) | 0 | 4
  Day 12: 24 hours post-dose |  | 90.5 (26.2)
  Day 25: pre-dose: number analyzed (Participants) | 4 | 0
  Day 25: pre-dose | 29.6 (6.05) |
  Day 25: 1 hour post-dose: number analyzed (Participants) | 4 | 0
  Day 25: 1 hour post-dose | 31.9 (10.8) |
  Day 25: 2 hours post-dose: number analyzed (Participants) | 4 | 0
  Day 25: 2 hours post-dose | 50.5 (21.2) |
  Day 25: 4 hours post-dose: number analyzed (Participants) | 4 | 0
  Day 25: 4 hours post-dose | 76.2 (21.9) |
  Day 25: 8 hours post-dose: number analyzed (Participants) | 4 | 0
  Day 25: 8 hours post-dose | 83.9 (29.4) |
  Day 25: 24 hours post-dose: number analyzed (Participants) | 4 | 0
  Day 25: 24 hours post-dose | 69.4 (20.4) |

23. Secondary Outcome: Phase 2a: Pharmacokinetics: Maximum Observed Plasma Concentration (Cmax) of Tesevatinib 150 mg
Description: Cmax was defined as maximum observed plasma concentration.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing
Number analyzed (Participants) | 5 | 5
ng/mL
  Day 1 | 56.1 (15.3) | 49.9 (20.3)
  Day 12: number analyzed (Participants) | 0 | 5
  Day 12 |  | 102 (41.5)
  Day 25: number analyzed (Participants) | 4 | 0
  Day 25 | 84.0 (29.2) |

24. Secondary Outcome: Phase 2a: Pharmacokinetics: Time of the Maximum Observed Plasma Concentration (Tmax) of Tesevatinib 150 mg
Description: Tmax was defined as time to reach maximum observed plasma concentration.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing
Number analyzed (Participants) | 5 | 5
hours
  Day 1 | 14.5 (8.84) | 7.20 (1.76)
  Day 12: number analyzed (Participants) | 0 | 5
  Day 12 |  | 12.0 (11.0)
  Day 25: number analyzed (Participants) | 4 | 0
  Day 25 | 7.03 (2.02) |

25. Secondary Outcome: Phase 2a: Pharmacokinetics: Time of the Last Quantifiable Plasma Concentration (Tlast) of Tesevatinib 150 mg
Description: Tlast was defined as time to reach last quantifiable plasma concentration.
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing
Number analyzed (Participants) | 5 | 5
hours
  Day 1 | 24.1 (0.163) | 20.8 (7.17)
  Day 12: number analyzed (Participants) | 0 | 5
  Day 12 |  | 20.0 (8.95)
  Day 25: number analyzed (Participants) | 4 | 0
  Day 25 | 24.2 (0.163) |

26. Secondary Outcome: Phase 2a: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time 0 to the Last Quantifiable Concentration (AUC0-t) of Tesevatinib 150 mg
Description: as for outcome 10
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing
Number analyzed (Participants) | 5 | 5
hr*ng/mL
  Day 1 | 1090 (274) | 866 (509)
  Day 12: number analyzed (Participants) | 0 | 5
  Day 12 |  | 1860 (1160)
  Day 25: number analyzed (Participants) | 4 | 0
  Day 25 | 1760 (559) |

27. Secondary Outcome: Phase 2a: Pharmacokinetics: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Post-dose (AUC0-24) of Tesevatinib 150 mg
Description: as for outcome 12
Time Frame: as for outcome 22
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing
Number analyzed (Participants) | 5 | 5
hr*ng/mL
  Day 1: number analyzed (Participants) | 5 | 4
  Day 1 | 1090 (277) | 1020 (424)
  Day 12: number analyzed (Participants) | 0 | 4
  Day 12 |  | 2280 (791)
  Day 25: number analyzed (Participants) | 4 | 0
  Day 25 | 1740 (551) |

28. Secondary Outcome: Phase 2a: Pharmacokinetics: Concentration Immediately Before Dosing (Ctrough) of Tesevatinib 150 mg
Description: Ctrough was the plasma concentration observed at the time immediately before study drug administration.
Time Frame: Bi-weekly: Pre-dose on Days 8, 11, 18 and 25; pre-dose on Months 2, 3, 4, 5 and 6; Tri-weekly: pre-dose on Days 3, 5, 8 and 12
Population: as for outcome 22
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing
Number analyzed (Participants) | 5 | 5
ng/mL
  Day 3: Pre-dose: number analyzed (Participants) | 0 | 4
  Day 3: Pre-dose |  | 37.2 [21.4 to 76.0]
  Day 5: Pre-dose: number analyzed (Participants) | 0 | 4
  Day 5: Pre-dose |  | 57.6 [34.2 to 116]
  Day 8: Pre-dose: number analyzed (Participants) | 5 | 4
  Day 8: Pre-dose | 28.0 [19.3 to 39.7] | 57.3 [30.7 to 132]
  Day 11: Pre-dose: number analyzed (Participants) | 5 | 0
  Day 11: Pre-dose | 38.8 [25.9 to 59.9] |
  Day 12: Pre-dose: number analyzed (Participants) | 0 | 5
  Day 12: Pre-dose |  | 53.7 [29.9 to 95.2]
  Day 18: Pre-dose: number analyzed (Participants) | 5 | 0
  Day 18: Pre-dose | 33.6 [15.2 to 43.3] |
  Day 25: Pre-dose: number analyzed (Participants) | 4 | 0
  Day 25: Pre-dose | 29.6 [20.6 to 33.9] |
  Month 2: Pre-dose: number analyzed (Participants) | 1 | 0
  Month 2: Pre-dose | 34.1 [34.1 to 34.1] |
  Month 3: Pre-dose: number analyzed (Participants) | 1 | 0
  Month 3: Pre-dose | 14.6 [14.6 to 14.6] |
  Month 4: Pre-dose: number analyzed (Participants) | 2 | 0
  Month 4: Pre-dose | 47.55 [38.2 to 56.9] |
  Month 5: Pre-dose: number analyzed (Participants) | 2 | 0
  Month 5: Pre-dose | 45.0 [25.4 to 64.6] |
  Month 6: Pre-dose: number analyzed (Participants) | 1 | 0
  Month 6: Pre-dose | 21.6 [21.6 to 21.6] |

ADVERSE EVENTS:
Time Frame: Phase 1b: From Baseline (Day 1) until 30 days after the last dose of study drug (i.e., up to 37 months) and Phase 2a: From Baseline (Day 1) until 30 days after the last dose of study drug (i.e., up to 29 months)
Description: Reported AEs were AEs that developed or worsened or became serious from the first dose (Day 1) of the study drug until 30 days after the last dose of study drug. Analysis was performed on safety population.
Arm/Group | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/8 | 0/5 | 0/10 | 0/14 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/8 | 0/5 | 1/10 | 0/14 | 1/8
Other Adverse Events (participants affected / at risk) | 24/24 | 8/8 | 5/5 | 10/10 | 14/14 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing (N=24) | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing (N=8) | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing (N=5) | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing (N=10) | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing (N=14) | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing (N=8)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b: Cohort 1: Tesevatinib 50 mg Once Daily Dosing (N=24) | Phase 1b: Cohort 2: Tesevatinib 100 mg Once Daily Dosing (N=8) | Phase 1b: Cohort 3: Tesevatinib 150 mg Once Daily Dosing (N=5) | Phase 2a: Cohort 4: Tesevatinib: Bi-weekly Dosing (N=10) | Phase 2a: Cohort 5: Tesevatinib: Tri-weekly Dosing (N=14) | Phase 2a: SILK Cohort: Tesevatinib 50 mg Once Daily Dosing (N=8)
Diarrhoea (Gastrointestinal disorders) | 10 | 4 | 2 | 5 | 6 | 2
Nausea (Gastrointestinal disorders) | 10 | 2 | 2 | 2 | 5 | 1
Vomiting (Gastrointestinal disorders) | 5 | 2 | 0 | 3 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 7 | 3 | 0 | 4 | 5 | 1
Blood creatinine increased (Investigations) | 4 | 3 | 1 | 1 | 2 | 2
Alanine aminotransferase increased (Investigations) | 4 | 2 | 0 | 2 | 1 | 2
Amylase increased (Investigations) | 4 | 0 | 0 | 0 | 5 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 2 | 0 | 2 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 2 | 0 | 1 | 1 | 0
Blood bicarbonate decreased (Investigations) | 3 | 0 | 0 | 0 | 2 | 0
Urine leukocyte esterase positive (Investigations) | 1 | 1 | 0 | 0 | 1 | 1
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 1
Bacterial test positive (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Blood urine present (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Cystatin C increased (Investigations) | 2 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Monocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Neutrophil count decreased (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | 0
Neutrophil count increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Blood bicarbonate increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood phosphorus increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Haematocrit increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Nitrite urine present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Protein total decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary sediment present (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Urine bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 8 | 4 | 4 | 1 | 3 | 0
Acne (Skin and subcutaneous tissue disorders) | 4 | 0 | 2 | 2 | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 0 | 0 | 2 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 2 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 0
Dry skin (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Urticaria (Investigations) | 1 | 0 | 0 | 1 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 6 | 1 | 1 | 1 | 5 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 3 | 2 | 1
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 1 | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 2 | 2
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 0 | 3 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 0
Conjunctivitis infective (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Streptococcal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Laryngitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0 | 0 | 5 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1 | 2 | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 0 | 0 | 2 | 3 | 1
Oedema peripheral (General disorders) | 1 | 1 | 1 | 1 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | 0
Pyrexia (General disorders) | 2 | 0 | 0 | 0 | 0 | 0
Infusion site rash (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 8 | 0 | 0 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 2 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 2 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 4 | 0 | 2 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 1 | 1
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 2 | 0
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Renal cyst ruptured (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Urine abnormality (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Urine odour abnormal (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 2
Sunburn (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | 0
Heat stroke (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Post procedural constipation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 4 | 0 | 0 | 1 | 2 | 3
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vitamin C deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 1 | 3 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 1 | 0
Mood altered (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Personality change (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 2 | 0 | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cystocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Polymenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Prostatic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectocele (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Uterine spasm (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 0 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 3 | 0 | 0 | 0 | 1 | 0
Eye discharge (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eye swelling (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lymphocyte count increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/63/NCT01559363/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/63/NCT01559363/SAP_001.pdf